CLINICAL TRIAL: NCT04971993
Title: Step and Walking Pattern From Cardiac Monitor Study
Acronym: SWAN
Status: Terminated | Type: Observational
Why Stopped: Resourcing challenges
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: C2168
Record Dates: First submitted 2021-06-28; First posted 2021-07-22 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III; Insertable Cardiac Monitor
Keywords: exercise; walk
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Heart Failure NYHA Class II: Participants are diagnosed with NYHA Class II heart failure.
  Interventions: Device: Wearable Cardiac Monitor
- Heart Failure NYHA Class III: Participants are diagnosed with NYHA Class III heart failure.
  Interventions: Device: Wearable Cardiac Monitor
- At risk for arrythmias: Participants are indicated for an insertable cardiac monitor with no history of heart failure.
  Interventions: Device: Wearable Cardiac Monitor

INTERVENTIONS:
Device: Wearable Cardiac Monitor — Participants will be fitted with a wearable cardiac monitor placed on their skin that measures physiological signals.

SUMMARY:
To understand the feasibility of characterizing walking patterns in heart failure subjects and subjects at risk for arrhythmias using an investigational wearable monitor called the SWAN study system.

DETAILED DESCRIPTION:
This is a non-randomized, feasibility study that will enroll up to 60 participants diagnosed with Class II (30-35%) or III (30-35%) heart failure or are indicated for an insertable cardiac monitor with no history of heart failure (30-35%).

There will be one study visit per participant and a follow up phone call. The study visit includes device placement and data collection during rest and during a 6 minute hall walk. The device will then be removed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older
* Willing and capable to provide written informed consent and agrees to participate in all protocol required activities
* Subjects must meet one of the following criteria:
* Documented New York Heart Association (NYHA) class II or III heart failure within the last 6 months

OR

* Subjects that have a known heart condition (non-heart failure) and are at risk of developing an abnormal heart rhythm, or have symptoms that may suggest a cardiac arrhythmia such as dizziness, palpitations, syncope, chest pain and/or shortness of breath

Exclusion Criteria:

* Not able to walk continuously for a period of 6 minutes at the subjects baseline walking speed
* Prior hospitalization or surgery that affects the subjects baseline walking speed at time of enrollment
* Cardiovascular event such as unstable angina or myocardial infarction that affects the subjects baseline walking speed at time of enrollment
* Subject is currently enrolled in another clinical trial (excluding registries) that may interfere with the placement of the study system
* Known allergy to materials used in the study (adhesive tape, titanium, ECG electrodes)
* Subject is pregnant as indicated by subject report and/or medical record at the time of enrollment
* Subjects with rash or open wound on torso locations where investigational devices will be placed
* Have an active implantable device
* Any past or current medical event that could represent a risk for the subject to perform the study required activities in the opinion of the investigator
* Any medical signs or symptoms that in the opinion of the investigator could represent a risk for the subject (I.e. increased baseline blood pressure or heart rate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are diagnosed with NYHA class II heart failure, class III heart failure or are indicated for an ICM with no history of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Step Detection | 12 months
  Characterize step count in class II and III heart failure and in ICM indicated patients with no history of heart failure.
Walking Patterns | 12 months
  Characterize walking patterns in class II and III heart failure and in ICM indicated patients with no history of heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Pelzel, MD, Principal Investigator — CentraCare Heart and Vascular Clinic
Locations (1):
- CentraCare Heart and Vascular Clinic, Saint Cloud, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No